CLINICAL TRIAL: NCT03265444
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of Autologous Bone Marrow Derived Mesenchymal Stem Cells in Subjects with Multiple System Atrophy
Brief Title: Safety and Tolerability of CS10BR05 Inj. in Subjects with Multiple System Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corestemchemon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS10BR05-MSA101
Record Dates: First submitted 2017-08-06; First posted 2017-08-29 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2020-08

CONDITIONS: Multiple System Atrophy
Keywords: MSA
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CS10BR05 (Experimental): The single injection of CS10BR05 Inj. in the carotid artery
  Interventions: Biological: CS10BR05

INTERVENTIONS:
Biological: CS10BR05 — The single injection of CS10BR05 Inj. in the carotid artery; Step 1 dose : 3.0x105cells/kg; Step 2 dose : 6.0x105cells/kg; Step 3 dose : 9.0x105cells/kg; The duration of follow up study following the single dose of CS10BR05 is 28 days.

SUMMARY:
The purpose of conducting phase 1 trial is to evaluate the safety and tolerability of autologous bone marrow-derived mesenchymal stem cells(CS10BR05) in subjects with Multiple System Atrophy.

Evaluation of DLT by carotid artery(intra-arterial) injection according to dose-escalating in Multiple System Atrophy.

DETAILED DESCRIPTION:
Multiple system atrophy is a neurodegenerative disease of the central nervous system which is accompanied by signs of autonomic imbalance (orthostatic hypotension, urinary problems, erectile dysfunction), Parkinson's symptoms (movement decreases, limb tremors) and cerebellar ataxia symptoms (grogginess, pronounced incorrectly). It shows signs similar to Parkinson's disease, however, it doesn't show improvement of symptoms by dopaminergic drugs and occurs at any age.

The clinical trial was designed as a single center, open-label, public phase 1 clinical trials.

If that subject's written consent to participate in this clinical trial will be conducted the required examinations and tests in accordance with the study protocol.

Then, the register for each dose step. For the final 3 subjects in the inclusion / exclusion criteria and be administered a drug test.

And check the adverse events for more than four hours after administration of the investigational drug, and will determine whether the expression of adverse drug reaction(ADR) by the visit after 1 days, 14 days and 28 days.

Except for dose administration, all subject are tested in the same schedule. As a result of evaluating severity of AE divided into subjective, objective in accordance with the CTCAE (Version 4.0) standards.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients aged ≥30 years and ≤ 75 years
* Meet criteria for diagnosis of probable MSA -cerebellar type according to the Gilman Criteria(2008)
* MRI or PET imaging showed a decrease in the cerebellar atrophy or cerebral metabolism
* Patients who are less than 4 years from the time of documented MSA diagnosis
* Patients unified MSA rating scale 30~50
* Those who have no hematologic abnormalities and who are not suspected of failing bone marrow function
* Patients who consented to participate in the study in writing by themselves or their legal representatives

Exclusion Criteria:

* Suspected clear Dementia (K-MMSE < 24)
* DSM-IV criteria for Dementia
* Radiologic imaging findings suggest that vascular encephalopathy coexist
* Other central nervous system diseases except MSA (Parkinsons disease etc.)
* Patients with Stroke or Brain surgery
* If there is a coexistence of severe medical illness, or if it is in a severe pyrexia state
* Serum SGOT / SGPT measures above three times of upper limit of normal or creatine levels were above 1.5 times of upper limit of normal levels were more than 1.5 times normal
* disease that affects the patient's long-term survival(Tumor, Serious Heart failure)
* Patients with genetic tests showed that spinocerebellar ataxia 1, 2, 3, 6, 7, 17
* Patients with unstable vital signs
* Patients with uncontrolled comorbidities such as moderate to severe infections, bleeding
* Those who are found to be active to viral infection(HBV, HCV, HIV, CMV, HTLVⅠ/Ⅱ, VDRL)
* Patients who are hypersensitive to bovine protein or antibiotics such as penicillin and streptomycin
* Patients with difficult catheter insertion(bleeding disorder, artery hardening narrowness, Patients who are at risk of stroke in cerebral angiography)
* Patients with cardiovascular disease(for example, hypertension, myocardial infarction etc;)
* Severe disease uncontrolled (diabetes)
* Those who are using drug likely to affect bone marrow functions
* Pregnant women or nursing women
* Women of childbearing age and male who do not consent to use proper contraception to prevent his partner from being pregnant during participation in the study
* Now clinical trials treated with other drugs and in clinical trials the previous 4 weeks
* Subjects who by the investigator to make them ineligible for participation in this clinical study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity and Maximum Tolerated Dose of CS10BR05 Inj. | up to 28days
  To evaluate the safety and tolerability of CS10BR05 Inj. in patients with Multiple System Atrophy including determination of its Dose Limiting Toxicity (DLT) and Maximum Tolerated Dose (MTD).
Adverse events, frequency and rate of vitals sign, laboratory test, physical examination, ECG, etc. | up to 28days
  To evaluate the safety and tolerability of CS10BR05 Inj. in patients with Multiple System Atrophy.

SECONDARY OUTCOMES:
Unified Multiple System Atrophy Rating Scale(UMSARS) | -35days, 28days
  Part I (Historical review), part II (Motor examination scale), part III (Autonomic examination), part IV (Global disability scale) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Phil Hyu Lee, M.D., Principal Investigator — Yonsei University
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Corestem Inc. — http://www.corestem.com